CLINICAL TRIAL: NCT01977079
Title: Procalcitonin and Threatened Premature Delivery
Acronym: MAPPRO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CHD061-13
Record Dates: First submitted 2013-10-24; First posted 2013-11-06 (Estimated); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Pregnancy; Premature Delivery
Keywords: pregnancy; premature birth; procalcitonin
MeSH Terms: conditions — Premature Birth | interventions — Procalcitonin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Premature birth (Other): At the end of the study patients will be divided into two groups: "Premature delivery" versus "No premature delivery." Prematurity is defined as a birth before 37.
  In each group, the procalcitonin rate be estimated with a confidence interval of 95% and compared from a logistic regression.
  Interventions: Other: procalcitonin
- Not premature birth (Other): At the end of the study patients will be divided into two groups: "Premature delivery" versus "No premature delivery." Prematurity is defined as a birth before 37.
  In each group, the procalcitonin rate be estimated with a confidence interval of 95% and compared from a logistic regression.
  Interventions: Other: procalcitonin

INTERVENTIONS:
Other: procalcitonin

SUMMARY:
Among all patients hospitalized for Threatened Premature Delivery (TPD), the rate of premature birth (PB) before 37 weeks is about 42%, which reflects the inability to accurately identify patients at high risk of PB. Currently, no clinical or biological marker is recognized as the most reliable in predicting the real risk of AP in case of MAP.

The purpose of this study is to improve the knowledge of predictors of preterm delivery compared with conventional blood markers by estimating serum procalcitonin according to premature delivery or not in patients hospitalized for preterm labor .

ELIGIBILITY:
Inclusion Criteria:

* age > 18 year
* Ongoing pregnancy with a start date of pregnancy known and confirmed by an ultrasound of the 1st Quarter performed between 10 and 14 weeks with a measurement of the crown-rump length
* hospitalization for preterm labor between 24 and 36 weeks of gestation
* Intact membranes,
* not opposed to participate in the study

Exclusion Criteria:

* Pregnancy uncertain term (no early ultrasound)
* Pregnancy combining a condition that can interfere with the assays performed,
* Uterine malformation known
* Multiple pregnancy,
* Premature rupture of membranes,
* Chrorio-amnionitis,
* Fetal malformation known
* Strapping
* GB> 15000 and CRP> 10 mg / L,
* No affiliation to a social security scheme.
* Woman with a measure of legal protection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2013-12; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
procalcitonin rate | up to 48 hours
  Estimate serum procalcitonin according to premature or not in patients hospitalized for preterm labor.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume DUCARME, PH, Principal Investigator — Centre hospitalier départemental Vendée
Locations (1):
- Centre hospitalier départemental Vendée, La Roche-sur-Yon, France

REFERENCES:
- [Result] Ducarme G, Desroys du Roure F, Le Thuaut A, Grange J, Vital M, Dimet J. Efficacy of serum procalcitonin to predict spontaneous preterm birth in women with threatened preterm labour: a prospective observational study. BMC Pregnancy Childbirth. 2018 Mar 7;18(1):65. doi: 10.1186/s12884-018-1696-2. PMID 29514604